CLINICAL TRIAL: NCT02544256
Title: Mild Hypothermia During Intracranial Aneurysm Clipping: Effect on Brain Microcirculation and Postoperative Vasospasms in Patients With Ruptured Aneurysms
Brief Title: Mild Hypothermia During Intracranial Aneurysm Clipping
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: higher mortality in another published study
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Dostalova Vlasta, MD, PhD, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201507-S16P
Record Dates: First submitted 2015-08-27; First posted 2015-09-09 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Microcirculation; Mild Hypothermia, Induced; Subarachnoid Hemorrhage, Aneurysmal; Aneurysmal Clipping; Vasospasms
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mild hypothermia (Experimental): After induction to general anaesthesia the patients will be cooled to 33° C. Targeted body temperature 33,8° C - 34,8° will be maintained up to the end of microcirculation measurement after aneurysm clipping.
  Interventions: Procedure: Mild hypothermia
- Normothermia (No Intervention): The body temperature will be maintained in the range 35,8° C - 36,8° C.

INTERVENTIONS:
Procedure: Mild hypothermia — Mild hypothermia during surgical clipping of brain aneurysm will be reached by cooling to body temperature 33,8° C - 34,8° and this temperature maintained up to the end of microcirculation measurement after aneurysm clipping.
  Arms: Mild hypothermia

SUMMARY:
The purpose of this study is to determine whether mild hypothermia causes reduction of vasoconstriction in microcirculation after clipping of aneurysms, and affects the blood flow in small diameter arteries at operating site (ischemia-hyperemia) and occurrence of vasospasms during the period of 14 postoperative days measured by transcranial Doppler.

DETAILED DESCRIPTION:
Methods: All the patients meeting the study criteria will be randomized into two groups. Normothermia (NT) group : during the whole period of surgery the body temperature will be maintained in the range 35.8° C - 36.8° C. Hypothermia (HT) group: After induction to general anaesthesia the patients will be cooled to body temperature 33.8° C - 34.8° and this temperature maintained up to the end of microcirculation measurement after aneurysm clipping. Warming up of the patients will start immediately afterwards. The target temperature at the time of extubation will be over 36° C in both groups (one of the extubation criteria).

Specific management: No pharmacological sedation (premedication) will be given to the patients. Cooling/warming mattress/blanket (PlastiPad® Blanketrol® III Cincinnati Sub-Zero, USA) will be placed on the operating table. Induction to general anesthesia will be with propofol 2 mg/kg/b.w i.v. (with possible adjustment according to age and/or physical status of the patient) and atracurium 0,5 mg/kg/b.w. i.v. After orotracheal intubation, the esophageal temperature probe will be inserted (depth of insertion 25 cm from the nostril). Afterwards, the envelope with randomization will be opened by the anaesthesiologist.

In HT group, the targeted body temperature will be set to 33° C and a bolus of saline 250 ml cooled to 5° C will be administered.

In NT group, the targeted body temperature will be set to 36° C and a bolus of saline 250 ml warmed to 37° C using infusion heater will be administered.

Standard preparation for the surgery will continue afterwards (insertion of central venous catheter, arterial catheter, urinary catheter). After finishing the preparation (coming of the surgeon), the infusion of mannitol 15% at the dose 0,5 g/kg i.v. is started and set for the duration of 40 minutes. Monitoring: basic monitoring (SpO2, ECG, end-tidal carbon dioxide (EtCO2), NIBP) together with extended monitoring (invasive blood pressure, response entropy/state entropy (RE/SE), neuromuscular transmission module (NMT), surgical plethysmography index (SPI).

Anesthesia management: Desflurane anesthesia in O2/air mixture with concentration of oxygen (FiO2) 0.45 will be used with targeted concentrations of desflurane according to the age groups initially (to achieve end-tidal concentration of desflurane 6 V%, 5.5 V%, 5 V%, 4.5 V%, and 4 V% in age groups 18 - 30, 30 - 40, 40 - 55, 55 - 65, and over 65 years respectively), further adjustment will be done to keep target RE/SE 40-50 in the individual patient. Analgesia will be provided by bolus i.v. administration of remifentanil 80 ug before induction, followed by continuous administration 0.25 ug/kg/min initially with further stepwise adjustment according to SPI (3-5 ml/hour steps). Target analgesia according to SPI is defined as the initial figure of SPI recorded 5 minutes after induction plus 10 points. Figures of SPI exceeding for 1 minute the target figure indicate the need of increasing the rate of remifentanil infusion. Atracurium boluses will be used for muscle relaxation, NMT monitoring by train of four (TOF) will be done in 5 minute intervals, TOF count over 1 indicating need of further atracurium bolus. Starting from dura mater suture, no further boluses of atracurium will be given.

Hemodynamic stability: Systolic and mean arterial pressures are maintained in the range of ± 15% of usually measured BP for individual patient. Decrease of BP bellow this figure in the duration of at least 5 minutes is indication for continuous administration of noradrenaline. Nimodipine is administered continuously during the whole procedure, infusion rate is set at the ICU, no adjustments are indicated at the OR. Volume therapy is provided by continuous balanced isotonic crystalloid infusion 5 ml/kg/h.

Microcirculation measurement: After craniotomy, microcirculation will be measured by SDF probe at the labelled sites of the brain (edge of craniotomy and at the distance of 2 cm from aneurysm). After aneurysm clipping, the measurement will be repeated at the same sites.

Finishing anaesthesia: At the beginning of skin suture, the remifentanil infusion is stopped. After finishing the skin suture, the administration of desflurane is stopped and end-tidal control flush out of desflurane is activated.

Extubation criteria: consciousness Glasgow coma scale (E-2-3/V-1-3/M-6), normotension including noradrenaline administration in stable continuous dose, normocapnia, spontaneous ventilation with respiratory rate (RR) over 10/minute, tidal volume (TV) 4-6 ml/kg, preserved coughing reflex, SpO2 over 95% without/with O2 administration, normothermia over 36° C, train of four ratio over 92%.

ELIGIBILITY:
Inclusion Criteria:

* Acute subarachnoidal hemorrhage based on ruptured aneurysm
* Hunt and Hess scale 1-4
* Clipping up to 72 hours after the rupture

Exclusion Criteria:

* Known cryoglobulinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Changes in Sidestream Dark Field (SDF) imaging variables | 1 and 2 hours after skin incision
  brain microcirculation will be measured by sidestream-dark field imaging (SDF) probe

SECONDARY OUTCOMES:
Changes in diameter of small brain arteries at operating site | 1 and 2 hours after skin incision
  will be measured by SDF probe
Occurrence of vasospasms | within the first 14 days after surgery
  measured by transcranial Doppler

OTHER OUTCOMES:
Days of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Glasgow outcome score (GOS) on discharge | 2 weeks after operation

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD, PhD, Study Director — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia